CLINICAL TRIAL: NCT02865200
Title: The Effectiveness of Dry Needling and Classic Physiotherapy Programs in The Patients Suffering From Chronic Low Back Pain Caused by Lumbar Disc Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ender Angın, Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EasternMU
Record Dates: First submitted 2016-07-14; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Syndrome; Physical Activity; Quality of Life
Keywords: Nutrition; Public Health
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling Application (Experimental): Dry needling was performed on active and/or latent TPs at Gluteus Medius, Quadratus Lumborum, Multifidus, Erector Spinae muscles of the subjects in the study groups without applying any local anesthetic substance. The needles were applied with a 90º angle for Multifidus, Quadratus Lumborum and Gluteus Medius muscles; while they were applied with a 45º angle for Erector Spinae muscles. Thin stainless steel needles of 0.25x0.40 mm and 0.30x0.60 mm were applied in infiltration form on the TP through many points in conformity with the injection technique. The needles were kept on the body for 20 minutes and at the 10th minute, the needle was rolled and re-stimulation was enabled. The treatment was applied twice a week, which is equal to 6 sessions in total.
  Interventions: Other: Dry Needling Application
- Classic Physiotherapy Program (Experimental): Hot-pack was applied for 20 minutes. Burst TENS was applied on the lumbar regions of the cases of the control group paravertebrally with 4-electrode reusable silicone rubber. The dimensions of electrode is 5x5cm. Pulse width was set for 100 µsn, pulse frequency was set for 2 Hz, cycle time is set for 0.5 seconds and the amplitude was increased until visible muscle contraction was reached. If the muscle contraction is lost during the session, the amplitude was increased again. The period of treatment was 6 sessions in total with 25 minutes of each.
  Ultrasound was paravertebrally applied to the lower back regions of the subjects. The treatment was applied with 1 MHz frequency, 1.5 W/cm2 power, for 6 minutes a day, for 10 sessions in total with direct contact with the patient's skin.
  Interventions: Other: Classic Physiotherapy Program

INTERVENTIONS:
Other: Dry Needling Application — Dry needling was performed on active and/or latent TPs at Gluteus Medius, Quadratus Lumborum, Multifidus, Erector Spinae muscles of the subjects in the study groups without applying any local anesthetic substance. The needles were applied with a 90º angle for Multifidus, Quadratus Lumborum and Gluteus Medius muscles; while they were applied with a 45º angle for Erector Spinae muscles. Thin stainless steel needles of 0.25x0.40 mm and 0.30x0.60 mm were applied in infiltration form on the TP through many points in conformity with the injection technique.
  Arms: Dry Needling Application
Other: Classic Physiotherapy Program — Hot-pack was applied for 20 minutes. Burst TENS was applied on the lumbar regions of the cases of the control group paravertebrally with 4-electrode reusable silicone rubber. The dimensions of electrode is 5x5cm. Pulse width was set for 100 µsn, pulse frequency was set for 2 Hz, cycle time is set for 0.5 seconds and the amplitude was increased until visible muscle contraction was reached. If the muscle contraction is lost during the session, the amplitude was increased again.
  Ultrasound was paravertebrally applied to the lower back regions of the subjects. The treatment was applied with 1 MHz frequency, 1.5 W/cm2 power, for 6 minutes a day, for 10 sessions in total with direct contact with the patient's skin.
  Arms: Classic Physiotherapy Program

SUMMARY:
Aim: This study was planned for comparing physical activity levels, nutrition quality and quality of life of the individuals that are diagnosed with and without metabolic syndrome (MetS) and that live in the Turkish Republic of Northern Cyprus (TRNC).

Method: 1200 individuals in total, in which (n: 660) individuals diagnosed with MetS and (n:660) individuals not diagnosed with MetS, participated in this study. Socio-demographic characteristics of the individuals that participated the study were registered with a survey form. The long form of the International Physical Activity Questionnaire was used for determining physical activity levels of the individuals; whereas total numbers of daily steps were carried out with pedometer. The 14-item Mediterranean Diet Adherence Screener (MEDAS) was used for the assessment of dietary habits, Nottingham Health Profile (NHP) was used for the assessment of health-related qualities of life of individuals and Beck Depression Inventory (BDI) was used for the assessment of depression. In addition, biochemical analysis and anthropometric measurements of individuals were also taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients among the ages of 35-70,
* Suffering from LBP for at least 3 months,
* Diagnosed with LDH having at least 1 active trigger point that can be cooperated .

Exclusion Criteria:

* Those with LDH that show neurological symptom,
* Having any orthopaedic problem at lower extremity and lower back region,
* Having sacroiliac joint problem, diagnosed with lumbar spondylolisthesis,
* Having any neurologic, rheumatic, oncologic problem,
* Who received any physiotherapy program at least 6 months before, patients having any corticosteroid treatment or oral medication
* Those having needle phobia were not included in the trial.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain assessed using the Short Form of McGill Pain Questionnaire-Visual Analogue Scale | 2 weeks
  The Short Form of McGill Pain Questionnaire-Visual Analogue Scale (MPQ-SF-VAS) was used in order to determine the pain intensity that the investigators use as primary outcome measure in the investigators study.

IPD SHARING:
Plan to Share IPD: No